CLINICAL TRIAL: NCT05482542
Title: Optimal Conditioning Regimen Protocol for Autologous Hematopoietic Stem Cell Transplantation of Relapsing Remitting Multiple Sclerosis
Brief Title: Optimal Conditioning Regimen for Autologous Transplantation of Relapsing Remitting Multiple Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding for support staff
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-7874
Record Dates: First submitted 2022-07-12; First posted 2022-08-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Autologous Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide/ATG Conditioning Regimen (Other): Cyclophosphamide (200 mg /kg) / rabbit antithymocyte globulin (6.0 mg/kg)
  Interventions: Other: Autologous hematopoietic stem cell transplantation; Drug: Cyclophosphamide/ATG
- Cyclophosphamide/Rituximab Conditioning Regimen (Other): Cyclophosphamide (200 mg/kg) / rituximab (1000 mg).
  Interventions: Other: Autologous hematopoietic stem cell transplantation; Drug: Cyclophosphamide/Rituximab

INTERVENTIONS:
Other: Autologous hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation
Drug: Cyclophosphamide/ATG — Cyclophosphamide/ATG
  Arms: Cyclophosphamide/ATG Conditioning Regimen
Drug: Cyclophosphamide/Rituximab — Cyclophosphamide/Rituximab
  Arms: Cyclophosphamide/Rituximab Conditioning Regimen

SUMMARY:
This study is designed to compare two non-myeloablative conditioning regimens (combination of chemotherapy and immune specific proteins against immune cells) for relapsing remitting multiple sclerosis (RRMS). The two conditioning regimens are the most commonly used world wide in clinical practice for the treatment of multiple sclerosis (MS). The first investigational conditioning regimen is cyclophosphamide (chemotherapy) and rATG (rabbit anti-thymocyte globulin, a protein against immune cells). The second investigational conditioning regimen includes the same dose of cyclophosphamide (chemotherapy) and rituximab (a protein against immune cells). Both cyclophosphamide and either rATG or rituximab are given to kill immune cells that are thought to be causing MS, followed by return of one's own previously collected blood stem cells (autologous stem cell transplant) to hasten recovery. The goal of this study is to assess the difference of these treatments in terms of toxicity and efficacy.

DETAILED DESCRIPTION:
Autologous hematopoietic stem cell transplantation (HSCT) in patients with active relapsing remitting multiple sclerosis (RRMS) halts disease progression, improves neurologic disability and quality of life, and provides a prolonged drug-free remission. A "position paper" by neurologists and hematologists under the American Society of Transplant and Cellular Therapy (ASTCT) has recommended autologous HSCT as standard of care, clinical evidence available, for treatment-refractory relapsing MS with high risk of future disability. Similarly, the EBMT has recommended the use of HSCT as "standard or care" for patients with highly active RRMS failing at least one DMT. Currently, the optimal conditioning regimen in terms of safety and efficacy is unknown. Herein, we will compare the two most commonly used regimens cyclophosphamide/ATG, or cyclophosphamide/rituximab in terms of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-58 years old
2. MRI T2 hyperintense lesions with at least 1 lesion in two or more of the following locations: periventricular, cortical or juxtacortical, infratentorial, or 1 spinal lesion
3. Since diagnosis a new MRI T2 lesion or since diagnosis a gadolinium positive lesion and at least one T2 weighted lesion
4. RRMS with a history of:

   1. 2 or more "active flares" in the prior 12 months despite either copaxone or interferon; or
   2. 1 or more "active flares" in the prior year despite a 2nd or 3rd generation DMT; or
   3. Active secondary progressive MS (aSPMS) with 2 or more gadolinium enhancing lesions with at least 1 gadolinium enhancing lesion > 5 mm in longest dimension within the last 9 months

Exclusion Criteria:

1. CIS- clinically isolated lesion
2. isolated optic neuritis
3. Primary progressive MS b) Nonactive SPSM (defined as no new or enhancing lesions in last 12 months)
4. spasticity or clinical stiffness of leg(s) unless there is documented new MRI enhancement within the past 12 months.
5. hyperreflexia or clonus
6. other immune neurologic disease such as NMO, CIDP, Stiff person syndrome, myasthenia gravis
7. genetic neurologic diseases such as CMT or spinal cerebellar degeneration
8. another autoimmune diagnosis such as systemic lupus erythematosus, systemic sclerosis, Behcets, or crohn's disease, etc (with the exception of hypo or hyperthyroidism or history of ITP or AIHA that is in remission)
9. insulin dependent diabetes mellitus
10. sickle cell disease
11. thalassemia major
12. porphyria
13. a current or prior cancer / malignancy except for cutaneous basal cell carcinoma or carcinoma in situ (completely excised)
14. Hepatic:

    1. Liver function test (AST or ALT) > 2 x upper limit of normal or
    2. bilirubin > 2.0 mg /dl
15. Pulmonary:

    1. DLCO < 60% of normal or;
    2. Asthma not easily corrected with bronchodilator therapy or;
    3. Pulmonary artery hypertension (pulmonary artery systolic pressure (PASP) > 40 mmHg on echocardiogram or by cardiac catheterization a mean pulmonary artery pressure (mPAP) > 25 mmHg; a cardiac catheterization for pulmonary artery pressures is only performed if clinically indicated)
16. Renal:

    1. creatinine > 2.0 mg/dl, or
    2. nephrotic syndrome
17. Cardiac:

    1. Acute myocardial infarction (AMI) within the last year, and if history of AMI not being approved by cardiology as low risk or not at increased risk for another AMI: or
    2. Persistent arrythmia not controlled with medication;
    3. Any patient requiring medication for an arrhythmia must be pre-approved by cardiology, or
    4. left ventricular ejection fraction < 45%
18. Hematology

    1. Hereditary coagulopathy or currently receiving anticoagulation therapy
    2. platelets < 100,000
    3. myelodysplastic syndrome
19. Infection:

    1. HIV,
    2. hepatitis B
    3. hepatitis C
    4. positive quantiferon gold (tuberculosis test) (may start HSCt once seen by ID and started on anti-tuberculous therapy, that will be continued throughout transplant, if asymptomatic),

    d) active infection at time of hospital admission (except UTI)
20. EDSS < 2.0 at time of enrollment or insurance submission
21. Inability to comprehend or give or sign informed consent
22. Pregnancy (positive serum or urine HCG test) or breast feeding
23. Failure to comprehend infertility as a complication.
24. Failure to offer sperm or oocyte collection and storage
25. Before HSCT failure to be Free of alemtuzumab for 12 months
26. Before HSCT failure to be Free of natalizumab for 5 months
27. Before HSCT failure to be Free of rituximab or ocrelizumab for 5 months
28. Before HSCT failure to be Free of fingolimod for 3 months
29. Before HSCT failure to be Free of dimethyl fumarate (tecfidera) for 3 months
30. Before HSCT failure of teriflunomide to have plasma levels < 0.02 mg/L after either oral cholestyramine or activated charcoal clearance.
31. Prior mitoxantrone
32. Prior cladribine

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Durability of remission between two arms | Time to first confirmed acute relapse or 5 years after treatment which ever comes first
  Defined as the time to first confirmed acute relapse or 5 years after treatment which ever comes first

SECONDARY OUTCOMES:
Neurologic Disability | From initiation of study to completion, up until 5 years after treatment
  Defined by change in EDSS (Expanded Disability Status Scale, ranges from 0 to 10 with 0 normal and 10 worst)

CONTACTS AND LOCATIONS:
Overall Officials: David J Hermel, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States